CLINICAL TRIAL: NCT07091994
Title: A Prospective, Multicentre, Randomized Controlled Trial of Edaravone Dexborneol in Acute Ischemic Stroke With Active Malignancy
Acronym: PRECISE AM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2025-303
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke, Acute; Active Malignancies
Keywords: active malignancies; ischemic stroke, acute; edaravone dexborneol; neuroprotection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This multicenter, randomized, open-label, controlled clinical trial will evaluate the efficacy and safety of edaravone dexborneol injection in patients with acute ischemic stroke (AIS) complicated by active malignancies. Eligible participants will be randomly assigned to receive either standard therapy combined with edaravone dexborneol injection or standard therapy alone for a treatment period of 10-14 days, followed by a 90-day follow-up period with scheduled assessments. The study will compare neurological functional recovery and safety profiles between the two treatment arms.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects randomized to the trial group will receive edaravone dexborneol injection at a dose of 37.5 mg (consisting of 30 mg edaravone and 7.5 mg dexborneol) administered twice daily with a fixed 12-hour interval between doses. The study drug will be diluted in 100 mL of normal saline and delivered via intravenous infusion over 30 minutes. This treatment regimen will be maintained for a duration of 10 to 14 days, in addition to standard stroke care. Strict adherence to the dosing schedule and infusion protocol will be ensured to maintain treatment consistency across study sites.
  Interventions: Drug: edaravone dexborneol injection; Drug: Standard therapeutic protocol
- Control group (Active Comparator): Subjects randomized to the control group will receive conventional standard therapy for acute ischemic stroke without the addition of edaravone dexborneol. The standard treatment regimen, which may include antiplatelet therapy, anticoagulation (if indicated), blood pressure management, and other evidence-based interventions, will be administered continuously for 10 to 14 days according to current clinical guidelines. All patients in this group will receive the same intensity of monitoring and follow-up as the experimental group to ensure comparable assessment of outcomes.
  Interventions: Drug: Standard therapeutic protocol

INTERVENTIONS:
Drug: edaravone dexborneol injection — The experimental intervention involved twice-daily administration of edaravone dexborneol injection at a dose of 37.5 mg (containing 30 mg edaravone and 7.5 mg dexborneol), with doses spaced exactly 12 hours apart. For each infusion, the study medication was first diluted in 100 mL of normal saline (0.9% sodium chloride solution) and then administered as a controlled intravenous infusion over a precisely timed 30-minute period. This standardized dosing regimen was maintained consistently throughout the 10-14 day treatment course for all participants in the experimental group.
  Arms: Intervention group
Drug: Standard therapeutic protocol — The standard treatment regimen, which may include antiplatelet therapy, anticoagulation (if indicated), blood pressure management, and other evidence-based interventions, will be administered continuously for 10 to 14 days according to current clinical guidelines.

SUMMARY:
This multicenter randomized controlled trial aims to evaluate the efficacy and safety of edaravone dexborneol injection in patients with acute ischemic stroke (AIS) complicated by active malignancies. The study will primarily investigate whether this combined antioxidant and anti-inflammatory treatment can improve neurological functional recovery and assess its safety profile in this high-risk population. Researchers will compare outcomes between the edaravone dexborneol treatment group and a control group receiving standard therapy to determine if the intervention provides superior neuroprotective effects. Participants will receive the assigned treatment regimen, undergo serial neurological assessments and imaging studies to monitor stroke progression and recovery, and be closely followed for safety evaluations. The findings may offer evidence-based therapeutic options for managing this challenging clinical scenario where current treatment alternatives are limited.

DETAILED DESCRIPTION:
Patients with acute ischemic stroke (AIS) who also have active malignancies face a more complex clinical scenario, with limited treatment options and generally poor prognoses. The coexistence of these two conditions can interact through inflammatory and oxidative stress pathways, forming a vicious cycle that exacerbates the patient's condition. Edaravone dexborneol injection exhibits significant antioxidant and anti-inflammatory effects, effectively scavenging free radicals in the body, thereby potentially improving the outcomes of AIS patients. Our team's preliminary retrospective study demonstrated that edaravone dexborneol injection can promote neurological recovery in AIS patients with active malignancies and shows a favorable safety profile. Therefore, this study aims to conduct a multicenter randomized controlled trial to evaluate the efficacy and safety of edaravone dexborneol injection in treating AIS patients with active malignancies, with the goal of providing evidence-based medical support and more effective therapeutic strategies for this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 80 years (inclusive); 2. Diagnosis of acute ischemic stroke (AIS) according to the 2023 Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke; 3. Time from symptom onset to enrollment ≤48 hours; 4. Presence of focal neurological deficits with a baseline NIHSS score of 4-24, and a combined score of ≥2 points on NIHSS Item 5 (upper limb motor) and Item 6 (lower limb motor); 5. Confirmed active malignancy before stroke onset or during hospitalization, defined as: Cancer diagnosed within 12 months prior to stroke, Presence of metastatic disease, Received cancer-directed therapy within the past 30 days, or Patients who declined cancer treatment (still considered active malignancy); 6. Signed informed consent obtained from the patient or legally authorized representative.

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded: 1. Intracranial hemorrhagic diseases detected on head CT: hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc; 2. Pre-stroke modified Rankin Scale (mRS) score >1; 3. Transient ischemic attack (TIA) as the current event; 4. Non-invasive skin cancers (e.g., basal cell carcinoma), primary central nervous system tumors, or hematologic malignancies; 5. Use of neuroprotective agents, including but not limited to: marketed edaravone, nimodipine, gangliosides, citicoline, piracetam, butylphthalide, human urinary kallidinogenase, or certain Chinese herbal medicines (see Concomitant Medications for details); 6. Patients with severe psychiatric disorders or dementia; 7.Hepatic or renal dysfunction: ALT or AST >3× upper limit of normal (ULN); Known liver diseases (e.g., acute/chronic active hepatitis, cirrhosis); Known kidney disease, renal insufficiency, serum creatinine >1.5×ULN, or creatinine clearance <50 mL/min; 8.Severe systemic diseases with an expected survival <90 days; 9. Pre-stroke Eastern Cooperative Oncology Group (ECOG) performance status ≥3; 10. Hypersensitivity to edaravone, (+)-borneol, or any excipients; 11. Pregnancy, lactation, or planned pregnancy; 12. Participation in another clinical trial within 30 days prior to randomization or current enrollment in other interventional studies; 13.Any other condition deemed inappropriate for participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in NIHSS score from baseline to Day 30 post-treatment. | From enrollment to the end of treatment at Day 30

SECONDARY OUTCOMES:
mRS score | From enrollment to the end of treatment at Day 30 and Day 90
Proportion of patients with mRS score ≤2 | From enrollment to the end of treatment at Day 30 and Day 90
Change in NIHSS score | From enrollment to the end of treatment at Day 14 and Day 90
Incidence of symptomatic intracranial hemorrhage transformation | From enrollment to the end of treatment at 36-48 hours and 7 days
Proportion of patients with Barthel Index (BI) score ≥95 | From enrollment to the end of treatment at Day 14, Day 30, and Day 90
All-cause mortality rate | From enrollment to the end of treatment at Day 30 and Day 90
Changes in serum inflammatory markers and coagulation parameters | From enrollment to the end of treatment at Day 14 and Day 30
Overall incidence of adverse events (AEs) | From enrollment to the end of treatment at 90 days
Incidence of treatment-emergent adverse events (TEAEs) | From enrollment to the end of treatment at 90 days
Occurrence of significant adverse events | From enrollment to the end of treatment at 90 days
Incidence of serious adverse events (SAEs) | From enrollment to the end of treatment at 90 days
Abnormalities in clinical laboratory tests | From enrollment to the end of treatment at 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Baiyun, China

IPD SHARING:
Plan to Share IPD: No